CLINICAL TRIAL: NCT03658642
Title: Pragmatic Trial of User-centered Clinical Decision Support to Implement EMergency Department-initiated BuprenorphinE for Opioid Use Disorder
Brief Title: Clinical Decision Support to Implement ED-initiated Buprenorphine for OUD
Acronym: EMBED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of North Carolina (Other); University of Alabama at Birmingham (Other); Mayo Clinic (Other); The Cooper Health System (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC 2000023783; UG3DA047003 (NIH)
Record Dates: First submitted 2018-08-28; First posted 2018-09-05 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Clinical Decision Support; Buprenorphine; Opioid-use Disorder
Keywords: Opioid Use Disorder; Buprenorphine; Opioid-use Disorder; Health IT
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Parallel cluster randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Decision Support for BUP (Experimental): The Clinical Decision Support (CDS) will be available for clinician use for Emergency Department (ED)-initiated buprenorphine/naloxone (BUP) with referral for ongoing medication assisted treatment (MAT) if: ED chief complaint or urine drug screen indicate opioid use. The clinician will then be prompted to complete DSM-5 checklist for OUD. If DSM-5 OUD Score>5 and urine drug screen is positive for opioids, then the clinician is prompted to complete COWS scale. If COWS score >12, then the clinician is prompted to order BUP. Regardless of COWS score, the clinician will be prompted to schedule an MAT appointment with BUP provider. The CDS will interface with outside MAT facilities so that making an appointment is easy and to capture data on whether an appointment has been scheduled.
  Interventions: Behavioral: Clinical Decision Support (CDS)
- Usual Care (No Intervention): The CDS will not be activated and patients will receive care as usual.

INTERVENTIONS:
Behavioral: Clinical Decision Support (CDS) — This clinical decision support tool will improve the clinician's ability to identify those with OUD, initiate BUP and refer the patient to ongoing Medication Assisted Treatment (MAT)
  Arms: Clinical Decision Support for BUP

SUMMARY:
Emergency Departments (EDs) frequently care for individuals with Opioid Use Disorder (OUD). Buprenorphine (BUP) is an effective treatment option for patients with OUD that can safely be initiated in the ED. At present, BUP is rarely initiated as a part of routine ED care. Clinical decision support (CDS) represents a potential approach to accelerate adoption of this best practice into routine emergency care. The goal of this trial is to determine whether implementation of a user-centered clinical decision support (CDS) system can increase adoption of initiation of BUP into the routine emergency care of individuals with OUD.

DETAILED DESCRIPTION:
The study design is an 18-month pragmatic, parallel, cluster randomized, superiority trial using constrained randomization of clusters to arms. The unit of randomization (i.e. cluster) is the ED. EDs will be randomly allocated with an allocation ratio of 1:1. Adequate lead time will be allotted to install the intervention in the electronic health records (EHR) at all intervention sites--including a three month implementation and washout phase. The intervention will then begin at the same time across all sites with the CDS intervention fully implemented in the intervention sites' EHRs at the start of the trial. Clinicians at control sites will retain all control of their practice and practice as usual without the CDS intervention installed in their EHR.

Pragmatic trials study an intervention under the usual conditions in which it will be applied; as opposed to an explanatory trial which would test an intervention under ideal conditions. In cluster randomized trials, treatment intervention is allocated to clusters (i.e. groups of individuals) rather than individuals. This is done to manipulate the physical or social environment of the intervention when an individual intervention would likely result in contamination between intervention and control participants at the group level. The parallel cluster randomized design was chosen over a stepped wedge design due to the high likelihood of confounding by temporal trends from ongoing efforts to mitigate the opioid epidemic. A major challenge of the cluster randomized design is from potential confounding due to a limited number of heterogeneous groups. Constrained randomization offers a solution to this source of confounding by balancing key cluster-level prognostic factors across the study to avoid distorting estimates of treatment effect due to the confounding factors. This allocation technique more evenly distributes potential confounders between intervention arms by specifying the confounding factors, characterizing each cluster in terms of these factors, identifying a subset of randomization combinations of clusters that adequately balance confounding factors between intervention arms and randomly selecting one of these combinations as the allocation scheme. Potential confounders that will be used for this trial are: EHR vendor, ED annual volume, ED type (e.g., academic, community, urban, rural, etc), ratio of ED clinicians who have a waiver to prescribe BUP, current rate of ED BUP prescribing, resources in ED to facilitate management of patients with OUD, and willingness of staff to adopt the practice of ED-initiation of BUP.

Intervention:

The intervention for this study includes the user-centered CDS as well as education of ED clinicians practicing at all study sites.

The need for flexibility in the graphical user interface of the intervention resulted in the decision to develop the CDS as a web application. This provides the ability to access the tool both embedded within the EHR or directly over the Internet. The web application was developed as a single-page application (SPA) based on React JavaScript library. The CDS is a user-initiated, Substitutable Medical Applications and Reusable Technologies (SMART) on Fast Health Interoperability Resources (FHIR) application that streamlines a flow diagram of the clinical protocol for ED-initiated BUP.

The intervention's graphical user interface is an intuitive, simple layout presenting four care pathways in columns based on the patient's diagnosis of OUD, the severity of withdrawal, and readiness to start treatment. There is additional, optional decision support available for guidance to: 1) evaluate OUD severity based on diagnostic and statistical manual of mental disorders (DSM)-5 criteria, 2) assess withdrawal severity using the clinical opiate withdrawal scale (COWS) score, and 3) motivate patient willingness and readiness to initiate medications for opioid use disorder (MOUD) treatment with a brief motivational interview. These materials are also available to share with other members of the care team via a web address, text messaging, or Quick Response (QR) code. The interface also includes a toggle switch for the user based on whether or not they have a waiver to prescribe BUP. Clinicians without a waiver cannot prescribe BUP but can administer a one-time dose of BUP in the ED for up to 72-hours. When integrated into the local EHR system, launching a care pathway enables the user to: place orders, refer for ongoing MOUD treatment, and update clinical notes.

The educational plan will be site-specific and tailored to the usual care at that institution. It will be administered within three months of the study start date. The details of the plan will be developed in partnership with local champions who self-identify an interest in helping to implement an ED-initiated BUP protocol at their site. Specifically, the education plan will be required to include:

1) A didactic on opioid use disorder, its diagnosis, assessment of withdrawal severity, and local resources for referral for ongoing MOUD treatment, 2)Circulation and posting in each study site ED of the flow diagram of the study's clinical protocol for ED-initiated BUP. Since this protocol is considered best practice, clinicians at control sites will retain all control of their practice and be encouraged to follow this protocol even though the CDS will not be available to them. 3) Intervention sites will include strategies to increase use of the intervention by training clinicians on how to launch and use the CDS. Use of the intervention will be tracked with site-specific audit and feedback that is consistent with typical quality improvement initiatives at that site.

Given the ongoing and escalating opioid epidemic and wide scope of this trial, the investigators anticipate that there may be concomitant interventions to stem OUD at study sites during the trial. The investigators plan to permit these interventions as long as they are: (1) implemented before randomization so that they can be tracked and accounted for in the constrained randomization process, and (2) they are not a health IT intervention targeted at clinicians to initiate BUP in the ED.

ELIGIBILITY:
Inclusion Criteria:

Clinicians

* All clinicians working in Emergency Departments in the selected sites

Patients

* 18 years or older
* Will meet an EHR-derived phenotype suggesting possible OUD will be included in the analysis
* Will be discharged from the ED
* Not pregnant
* Not currently taking any medication for Opioid Use Disorder

Exclusion Criteria:

Patients

* Have a medical or psychiatric condition that requires hospitalization during the ED visit
* Have prior enrollment in the current study
* Currently in addiction treatment
* Be a prisoner or in police custody at the time of ED visit

Note: The CDS will also be available for physicians to use when patients do not meet the EHR phenotype. These patients will be excluded from the primary analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5047 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Melnick, MD, MHS, Principal Investigator — Yale University
Locations (22):
- United States (22):
  - UAB Medicine Highlands - Highlands ED, (HED), Birmingham, Alabama
  - UAB - University Hospital ED (UED), Birmingham, Alabama
  - UAB Freestanding Emergency Department of Gardendale (GED), Gardendale, Alabama
  - UCHealth Anschutz Medical Campus (AMC), Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - UCHealth Memorial Hospital North (MHN), Colorado Springs, Colorado
  - UCHealth Poudre Valley Hospital (PVH), Fort Collins, Colorado
  - UCHealth Medical Center of the Rockies, Loveland, Colorado
  - Bridgeport Hospital ED (BPT), YNHHS, Bridgeport, Connecticut
  - Greenwich Hospital ED (GH), YNHHS, Greenwich, Connecticut
  - St Raphael's Campus (SRC), YNHHS, New Haven, Connecticut
  - Lawrence + Memorial Hospital ED (L&M), YNHHS, New London, Connecticut
  - Baystate Franklin, Greenfield, Massachusetts
  - Baystate Wing Hospital ED, Palmer, Massachusetts
  - Baystate Springfield Hospital ED, Springfield, Massachusetts
  - Baystate Mary Lane Hospital ED, Ware, Massachusetts
  - Baystate Noble, Westfield, Massachusetts
  - UNC Hospitals Emergency Department, UNCHS, Chapel Hill, North Carolina
  - REX Healthcare Emergency Department, UNCHS, Raleigh, North Carolina
  - Emergency Care Center at Nash General Hospital, UNCHS, Rocky Mount, North Carolina
  - Chatham Hospital ED, UNCHS, Siler City, North Carolina
  - Johnston Health ED, UNCHS, Smithfield, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cowan E, D'Onofrio G, Perrone J, Anderson E, Dziura J, Hawk K, Herring A, McCormack R, Phadke M, Samuels EA, Fiellin DA. Drug Use After Emergency Department-Initiated Injectable Buprenorphine: A Secondary Analysis of the ED-INNOVATION Ancillary Safety and Feasibility Trial. Acad Emerg Med. 2025 Nov 24. doi: 10.1111/acem.70191. Online ahead of print. PMID 41287157
- [Derived] Gao E, Melnick ER, Paek H, Nath B, Taylor RA, Loza AJ. Adoption of Emergency Department-Initiated Buprenorphine for Patients With Opioid Use Disorder: Secondary Analysis of a Cluster Randomized Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2342786. doi: 10.1001/jamanetworkopen.2023.42786. PMID 37948075
- [Derived] Melnick ER, Nath B, Dziura JD, Casey MF, Jeffery MM, Paek H, Soares WE 3rd, Hoppe JA, Rajeevan H, Li F, Skains RM, Walter LA, Patel MD, Chari SV, Platts-Mills TF, Hess EP, D'Onofrio G. User centered clinical decision support to implement initiation of buprenorphine for opioid use disorder in the emergency department: EMBED pragmatic cluster randomized controlled trial. BMJ. 2022 Jun 27;377:e069271. doi: 10.1136/bmj-2021-069271. PMID 35760423
- [Derived] Melnick ER, Nath B, Ahmed OM, Brandt C, Chartash D, Dziura JD, Hess EP, Holland WC, Hoppe JA, Jeffery MM, Katsovich L, Li F, Lu CC, Maciejewski K, Maleska M, Mao JA, Martel S, Michael S, Paek H, Patel MD, Platts-Mills TF, Rajeevan H, Ray JM, Skains RM, Soares WE 3rd, Deutsch A, Solad Y, D'Onofrio G. Progress Report on EMBED: A Pragmatic Trial of User-Centered Clinical Decision Support to Implement EMergency Department-Initiated BuprenorphinE for Opioid Use Disorder. J Psychiatr Brain Sci. 2020;5:e200003. doi: 10.20900/jpbs.20200003. Epub 2020 Feb 21. PMID 32309637
- [Derived] Melnick ER, Jeffery MM, Dziura JD, Mao JA, Hess EP, Platts-Mills TF, Solad Y, Paek H, Martel S, Patel MD, Bankowski L, Lu C, Brandt C, D'Onofrio G. User-centred clinical decision support to implement emergency department-initiated buprenorphine for opioid use disorder: protocol for the pragmatic group randomised EMBED trial. BMJ Open. 2019 May 30;9(5):e028488. doi: 10.1136/bmjopen-2018-028488. PMID 31152039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Physicians in the study were not "enrolled" but rather were found in the electronic health record data used in the study.
Period: Patients
Arm/Group | Clinical Decision Support for BUP | Usual Care
Started | 2787 | 2260
Completed | 2787 | 2260
Not Completed | 0 | 0
Period: Physicians
Arm/Group | Clinical Decision Support for BUP | Usual Care
Started | 340 (A total of 599 physicians were also included in the study.) | 259 (A total of 599 physicians were also included in the study.)
Completed | 340 | 259
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 5047 patients included in this study. The 599 physicians were not considered enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Decision Support for BUP | Usual Care | Total
Number analyzed (Participants) | 2787 | 2260 | 5047
Age, Categorical [Count of Participants; unit: Participants] — Categorical Age Grouping for Physicians Population: There were 599 physicians included in the study, 524 physicians (75 missing) had demographic information.
  Participants
    number analyzed (Participants) | 314 | 210 | 524
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 305 | 203 | 508
    >=65 years | 9 | 7 | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age, continuous for patients in the study.
  years | 36 [29 to 48] | 36 [29 to 46] | 36 [29 to 47]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5047 patients had demographic information, 524 physicians (75 missing) had demographic information.
  Participants
    Patients: Female | 917 | 813 | 1730
    Patients: Male | 1870 | 1447 | 3317
    Physician: number analyzed (Participants) | 314 | 210 | 524
    Physician: Female | 104 | 69 | 173
    Physician: Male | 210 | 141 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Race/Ethnicity was not collected for the physicians in the study.
  Participants
    Hispanic or Latino | 505 | 196 | 701
    Not Hispanic or Latino | 2166 | 1934 | 4100
    Unknown or Not Reported | 116 | 130 | 246
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race/Ethnicity was not collected for the physicians in the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 452 | 406 | 858
    White | 2048 | 1565 | 3613
    More than one race | 196 | 219 | 415
    Unknown or Not Reported | 91 | 70 | 161
Region of Enrollment [Number; unit: participants] — 5047 patients, 599 physicians combined.
  participants
    United States | 3127 | 2519 | 5646

OUTCOME MEASURES:

1. Primary Outcome: Count of Initiating BUP in the ED With Referral for Ongoing MOUD With User-centered CDS Compared With Usual Care
Description: The primary outcome will be Buprenorphine (BUP) initiation in the Emergency Department (ED), defined as whether or not an eligible patient is administered BUP in the ED and/or prescribed BUP upon discharge from the ED. Although this is not a patient-centered outcome, it is a pragmatic and meaningful surrogate that will serve as a lead indicator of the CDS intervention's effect on engaging more OUD patients in treatment. Medications for Opioid Use Disorder (MOUD)
Time Frame: Upon discharge (Up to 1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support for BUP | Usual Care
Number analyzed (Participants) | 2787 | 2260
Participants | 347 | 271
Statistical Analysis 1: Comparison: Clinical Decision Support for BUP vs Usual Care; Test type: Superiority; p = 0.58, GEE; Obtained from a GEE model accounting for clustering by site and multiple covariates; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.61 to 2.43]

2. Secondary Outcome: Count of Those With Referral to Follow-up for Ongoing MOUD Treatment (Patient Level)
Description: The count of enrolled patients who receive an Medication Assisted Therapy (MAT) appointment. Medications for Opioid Use Disorder (MOUD)
Time Frame: Upon discharge (Up to 1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support for BUP | Usual Care
Number analyzed (Participants) | 2787 | 2260
Participants | 367 | 226
Statistical Analysis 1: Comparison: Clinical Decision Support for BUP vs Usual Care; Test type: Superiority; p = 0.95, GEE; Obtained from a GEE model accounting for clustering by site; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.43 to 2.47]

3. Secondary Outcome: Rates Receiving a MAT Appointment Who go to the Appointment
Description: Data will be collected in the aggregate for the percentage of patients that attended the referral MAT appointment
Time Frame: 18 months
Population: These data were not able to be obtained.
Arm/Group | Clinical Decision Support for BUP | Usual Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Clinicians Providing ED-initiated BUP
Description: Number of clinicians providing ED-initiated BUP regardless of CDS
Time Frame: 18 months
Population: Clinicians participating in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support for BUP | Usual Care
Number analyzed (Participants) | 340 | 259
Participants | 151 | 88
Statistical Analysis 1: Comparison: Clinical Decision Support for BUP vs Usual Care; Test type: Superiority; p = 0.01, GEE; Obtained from a GEE model accounting for clustering by site; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.11 to 2.16]

5. Secondary Outcome: Number of Clinicians Providing Referral of Any Ongoing MOUD Treatment
Description: Number of clinicians that refer patients with OUD regardless of CDS
Time Frame: 18 months
Population: Clinicians participating in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support for BUP | Usual Care
Number analyzed (Participants) | 340 | 259
Participants | 141 | 100
Statistical Analysis 1: Comparison: Clinical Decision Support for BUP vs Usual Care; Test type: Superiority; p = 0.48, GEE; Obtained from a GEE model accounting for clustering by site; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.91 to 1.57]

6. Secondary Outcome: Number of Clinicians Who Have Received Drug Addiction Treatment Act (DATA) of 2000 Training
Description: Number of clinicians that obtained DATA waiver
Time Frame: 18 months
Population: Clinicians participating in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support for BUP | Usual Care
Number analyzed (Participants) | 340 | 259
Participants | 50 | 30
Statistical Analysis 1: Comparison: Clinical Decision Support for BUP vs Usual Care; Test type: Superiority; p = 0.27, GEE; Obtained from a GEE model accounting for clustering by site; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.81 to 2.14]

ADVERSE EVENTS:
Time Frame: 1 day
Description: Data for adverse events on patients would have been collected at the time of the encounter with the physician. Adverse events were not monitored or assessed in physicians.
Arm/Group | Clinical Decision Support for BUP | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/2787 | 0/2260
Serious Adverse Events (participants affected / at risk) | 0/2787 | 0/2260
Other Adverse Events (participants affected / at risk) | 0/2787 | 0/2260

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT03658642/Prot_SAP_000.pdf